CLINICAL TRIAL: NCT02490943
Title: A Pilot Study of Warm and Cold Compress to Reduce Injection Site Erythema Due to Peginterferon-beta-1a in Multiple Sclerosis
Brief Title: A Pilot Study of Warm and Cold Compress to Reduce Injection Site Erythema Due to Peginterferon-beta-1a in MS
Acronym: PEG-Thermal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown, Theodore R., M.D., MPH (Individual)
Collaborators: Evergreen Healthcare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TRB2015
Record Dates: First submitted 2015-06-24; First posted 2015-07-07 (Estimated); Last update posted 2022-03-25 (Actual); Status verified 2019-01

CONDITIONS: MS (Multiple Sclerosis); Erythema
Keywords: peginterferon beta-1a; MS (Multiple Sclerosis); Injection Site Reaction Erythema
MeSH Terms: conditions — Multiple Sclerosis; Erythema

STUDY DESIGN:
Intervention Model Description: Participants were randomized to warm compress (WC) for three injections, followed by cold compress (CC) for three injections, CC followed by WC, each for three injections or no treatment for six injections
Oversight: Data Monitoring Committee: No

ARMS (3):
- Warm Compress Pre-Injection (Active Comparator): Group A, N = 10, will receive warm compress before injection for three treatments, followed by cold compress after injection for three treatments.
  Interventions: Other: Warm Compress Before Injection
- Cold Compress Post-Injection (Active Comparator): Group B, N= 10, will receive cold compress after injection for three treatments followed by warm compress before injection for three treatments.
  Interventions: Other: Cold Compress After Injection
- No Intervention Pre/Post-Injection (No Intervention): Group C, N= 8, will receive no treatment for six injections following screening.

INTERVENTIONS:
Other: Warm Compress Before Injection — Receive warm compress before injection for three treatments, followed by cold compress after injection for three treatments.
  Other Names: Group A
  Arms: Warm Compress Pre-Injection
Other: Cold Compress After Injection — Receive cold compress after injection for three treatments followed by warm compress before injection for three treatments.
  Other Names: Group B
  Arms: Cold Compress Post-Injection

SUMMARY:
Peginterferon-beta-1a (PEG) is an approved treatment for relapsing forms of MS that may cause injection related erythema. This is a randomized controlled cross-over trial of superficial hot and cold modalities to reduce injection site erythema caused by PEG.

DETAILED DESCRIPTION:
The most common adverse event associated with this subcutaneously (SC) injected drug is injection site reaction (ISR) including redness and pain.Theoretically, both heat and cold modalities may improve interferon injection tolerance. Warm compress before injection may increase local blood flow and increase rapid systemic absorption, while cold compress afterward may reduce the erythema, edema and pain that often follow SC injections. A trial comparing heat-before and cold-after therapy is warranted to determine the relative effectiveness of these modalities.

Intervention:

Product: Reusable cold and warm compress.

Patients will receive written instructions for microwave heating and freezer cooling of the compress.

Warm compress: Pre-heating in microwave oven, per instructions. Apply warm compress for 5 minutes prior to injection. The initial compress temperature will be about 43 degrees Celsius (range 40-46 degrees Celsius) and slowly decline during application. Administer drug soon after removal.

Cold compress: Cooling in a freezer as per instructions. Soon after drug injection, apply cold compress for 10 minutes. The initial compress temperature will range 15-18 degrees Celsius.

* Timers will be utilized to mark 5-minute and 10-minute treatment intervals
* Participants will be encouraged to maintain constant practices with regards to non-steroidal anti-inflammatory drug use during the study

Study Objectives:

1. To assess and compare the impact on erythema of two thermal treatments: warm compress prior to PEG injection and cold compress following PEG injection
2. To assess the natural history of PEG-erythema over time. This will be accomplished with 18 weeks of observation in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS made at least 3 months prior based on McDonald criteria.
* Age 18 or more
* Ongoing treatment with PEG for 30 days or more at screening
* No MS exacerbation for 60 days prior to screening.
* Score of ≥50 on screening ISR Erythema Index
* Home access to microwave oven and freezer
* Written informed consent

Exclusion Criteria:

* Any contraindication to warm or cold compress:

  * Inability to sense temperature change by patient report
  * Metal implant near injection site (e.g. injection near intra-abdominal baclofen pump)
  * History of allergy or intolerance to local heat or cold application
  * Bleeding disorder
* Concomitant use of any topical prescription medication at injection site
* Females who are breast-feeding, pregnant or have potential to become pregnant during the course of the study (fertile and unwilling/unable to use effective contraceptive measures)
* Cognitive deficits that would interfere with the subject's ability to give informed consent or perform study testing.
* Any other serious and/or unstable medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-06; Primary Completion 2019-01-01 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline ISR Erythema Index at 24 hours, 7 days, and 14 days every 6 weeks for 18 weeks. | 24 hours, 7 days, 14 days
  Participants will record the diameter of patch of skin discoloration in millimeters, measuring at the maximum width.

SECONDARY OUTCOMES:
Change from baseline in rating of Modified Local Injection Site Reaction Scale | 24 hours
Erythema score on the Visual Assessment Scale. | Change from Baseline in VAS at 24 hours, 7 days, and 14 days.
  This is a 5 point visual assessment scale. Participants will be asked to observe the change in skin color at the site of injection. They will rate the intensity of skin color change (erythema) using the scale below. These assessments will be recorded at the following time points: 24 hours, 7 days, and 14 days
Pain score on the visual analogue scale after 10-minutes. | 10 min.
  (post-injection, 0-10 visual analogue scale (VAS))
Pain score on the visual analogue scale Post-Injection 24 hours, 7 days, and 14 days | Change from Baseline in VAS at 24 hours, 7 days, and 14 days.
  (post-injection, 0-10 visual analogue scale (VAS))
Level of Comfort Post-Injection Impression of Last 3 Weeks. | 18 Weeks
  This is a single question: "How would you rate your level of comfort with the last three injections?" This is on a 0-10 VAS with 0= "extremely bad" 5="neither good nor bad" and 10= "extremely good." The question will be answered at the end of each phase of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore R Brown, M.D., MPH, Principal Investigator — Evergreen Health Nueroscience Institute
Locations (1):
- Evergreen Health, Kirkland, Washington, United States